CLINICAL TRIAL: NCT03480997
Title: A Single Center Study to Measure the Bronchodilator Effect of Albuterol Sulfate or Albuterol Sulfate/Ipratropium Bromide Using the Pneuma Respiratory Inhaler and the ProAir HFA Inhaler in Stable COPD Patients
Brief Title: Acute Bronchodilator Effect of Inhaled Albuterol Sulfate and Ipratropium Bromide in Patients With Stable COPD
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pneuma Respiratory, Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2016-01
Record Dates: First submitted 2018-03-05; First posted 2018-03-29 (Actual); Last update posted 2018-03-29 (Actual); Status verified 2018-03

CONDITIONS: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Albuterol; Ipratropium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (3):
- albuterol sulfate 100 mcg (Experimental): albuterol sulfate 100 mcg Test MDI
  Interventions: Combination Product: Albuterol Sulfate
- albuterol sulfate 200 mcg (Active Comparator): albuterol sulfate 200 mcg Reference MDI
  Interventions: Combination Product: Albuterol Sulfate
- albuterol sulfate and ipratropium bromide (Experimental): albuterol sulfate 100 mcg and ipratropium bromide 20 mcg Test MDI
  Interventions: Combination Product: Albuterol Sulfate and Ipratropium Bromide

INTERVENTIONS:
Combination Product: Albuterol Sulfate and Ipratropium Bromide
  Arms: albuterol sulfate and ipratropium bromide
Combination Product: Albuterol Sulfate
  Arms: albuterol sulfate 100 mcg; albuterol sulfate 200 mcg

SUMMARY:
The purpose of this study is to demonstrate the pharmacodynamic bioequivalence of the test product to the reference product as measured by increases in FEV1.

DETAILED DESCRIPTION:
A single center, open label, single dose study to demonstrate the pharmacodynamic bioequivalence of the test and reference metered dose inhalers containing albuterol sulfate or albuterol sulfate/ipratropium in adult patients with COPD.

ELIGIBILITY:
Inclusion Criteria:

* Provide written informed consent
* Diagnosis of COPD as defined by the American Thoracic Society/European Respiratory Society guidelines characterized by progressive airflow limitation associated with abnormal inflammatory response of the lungs to noxious particles or gases primarily caused by cigarette smoking.
* Have an established COPD clinical history, symptomatic with dyspnea, chronic cough, chronic sputum production or wheezing. At Visit 1, FEV1/FVC ratio must be less than 0.70 or at least 10% less than the FEV1/FVC ratio determined by the predicted normal value. FEV1 must be less than 70% of the predicted normal value and greater than 25% of the predicted normal value.
* Must be using one or more inhaled bronchodilators for treatment of COPD at the time of Visit 1.
* Current or former smokers, with a history of at least 10 pack-years of cigarette smoking. Number of pack-years = (number of cigarettes per day/20) X (number of years smoked).
* Willing, and in the opinion of the investigator, able to adjust current COPD therapy as required by the protocol.

Exclusion Criteria:

* Current diagnosis of other respiratory disorder(s) including, but not limited to: alpha-1-antitrypsin deficiency; lung cancer; cystic fibrosis; tuberculosis; sarcoidosis; idiopathic pulmonary fibrosis; primary pulmonary hypertension; or pulmonary thromboembolic disease. Patients with concomitant COPD and asthma will be allowed to participate.
* Diagnosis of non-respiratory disorder(s) that are currently affecting lung function, as determined by he principal investigator including, but not limited to: congestive heart failure; symptomatic cardiac arrhythmia; symptomatic seizure disorder; dementia; lupus; rheumatoid arthritis; or liver cirrhosis.
* Unable to abstain from protocol defined prohibited medications during the screening and testing period.
* Unable to withhold short acting bronchodilators for 6 hours prior to spirometry testing at the study visit.
* Unable to perform acceptable or repeatable spirometry or comply with other study procedures.
* Known allergic reaction to albuterol sulfate or ipratropium bromide.
* Diagnosis of cancer that is not presumed to be in remission or cured.
* Active alcohol or drug abuse.
* Pregnant or lactating women. Pregnancy confirmed by a positive hCG test.
* Treatment with another investigational study drug in another clinical study within the last 30 days or five half-lives, whichever is longer.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2016-12-27 (Actual); Primary Completion 2017-04-28 (Actual); Study Completion 2017-04-28 (Actual)

PRIMARY OUTCOMES:
Primary Efficacy Endpoint: Change in FEV1 | Just prior to dosing and twenty minutes post dosing
  Change in FEV1

CONTACTS AND LOCATIONS:
Overall Officials: Tom Stern, MD, Principal Investigator — Advanced Respiratory and Sleep Medicine, PLLC
Locations (1):
- Advanced Respiratory and Sleep Medicine, PLLC, Hickory, North Carolina, United States